CLINICAL TRIAL: NCT06084429
Title: Developing School Health Champions to Increase Health Literacy Both in School Adolescents and Community People Through Providing Health Education by the School Nurses in Bangladesh: Community-based Pre- and Post-experimental Design.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Popi Rani Bhowmik, Doctoral Student, Hiroshima University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023/OR-NSU/IRB/0707
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Health Literacy
MeSH Terms: interventions — Lead

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pre and post test (Experimental): School adolescents studying in 8th grade.
  Interventions: Other: pre and post test (health educational intervention)

INTERVENTIONS:
Other: pre and post test (health educational intervention) — The health education will be provided the following sessions.
  Introduction to Global and Bangladesh Health, Health Information access (Validity), Critical Values (Vital signs, BMI, RBS etc.), Emergency Management (burn, chocking, knife cut, fainting etc.), Food (classification, healthy food, unhealthy, food label, salt intake) (NCDs from unhealthy diet), Smoking and Alcohol (NCD related, substance abuse, secondhand smoking), Physical activity (Benefits, sedentary lifestyle, NCD related), Women's health (menstruation, menstrual cycle, hygiene, STD, contraception), Hygiene (water, food, brushing, bath, toileting, healthy habits), Environmental Sanitation and Communicable disease (clean, effects on health), and Women's health and societal contribution

SUMMARY:
Health literacy is a person's decision-making ability to improve their quality of life and prevent diseases by accessing, understanding and applying health information. Health literacy in the adolescent's period can aid them to gain and understand health information which can bring positive health outcomes.

The aim of this pilot study is to examine the efficacy of health education and school health activities provided by school nurses on improving health literacy among secondary school adolescents. The study will also examine whether health education by health champions (the adolescents) is effective in improving the health literacy of the community people, and examine whether these interventions develop awareness, improve health knowledge, empower, and change behaviors of secondary school adolescents.

This intervention study aims to improve health literacy in the adolescents in Bangladesh and the school-located community. The Begum Ayesha Pilot Girl's High School in Dohar, Dhaka district will be selected as a field. First, we will place school nurses at the school, provide health checkups for both the adolescents (about n=316) and community people (about n=200), and school nurses will provide weekly health education for 3 months to the adolescents. After certifying them as "Health Champions", the health champions visit the community and provide health education activities to the community people. For both participant groups, health literacy will be measured as efficacy checking of this pilot study.

Assent and informed consent will be obtained from the participants. Autonomy, beneficence, non-maleficence, fidelity, veracity, confidentiality, and justice of the participants will be ensured. Also, anonymity will be maintained across all stages of the study.

ELIGIBILITY:
Inclusion Criteria:

For school adolescents:

* Students who are willing to participate.
* Students who study in class 8 (Grade 8) at the time of enrollment.
* Students who are female.
* Students whose parents or legal guardians agree to give consent and are willing to participate in the study
* Students who agree to receive health checkup, and are willing to respond to the questionnaire.
* Students who will stay in the same school till study completion.

For community people:

* Persons who are aged at least 18 years old.
* Persons who are willing to participate.
* Persons who agree to receive health checkup, and willing to respond to the questionnaire.
* Persons who will attend the health education activities.

Exclusion Criteria:

For school adolescents:

• Students who are absent from school during the health checkup periods due to severe illness or without any reason or information

For community people:

* Persons who will not attend the education sessions physically.
* Persons who will not live in the community until the post-test.

Ages: 11 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 138 (Actual)
Dates: Start 2024-02-24 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in health literacy score among the secondary school students | Baseline, Midline (after 3 months of baseline), Endline (after 6 months of baseline)
  Primary outcome will be measured by the health literacy scale for school-aged Children (HLSAC), Bangla version.

SECONDARY OUTCOMES:
Change in ratio of the level of health literacy | Baseline, Midline (after 3 months of baseline), Endline (after 6 months of baseline)
  This will be measured by HLSAC, Bangla version.
Change in self-efficacy score | Baseline, Midline (after 3 months of baseline), Endline (after 6 months of baseline)
  this will be measured by General Self-Efficacy Scale (GSE)
Change in reproductive age women specific health literacy | Baseline, Midline (after 3 months of baseline), Endline (after 6 months of baseline)
  This will be measured by using the Health literacy scale for women of reproductive age, Bangla version
Change in awareness and knowledge score | Baseline, Midline (after 3 months of baseline), Endline (after 6 months of baseline)
  This will be measured by the researcher-developed scale
Change in health behavior score | Baseline, Midline (after 3 months of baseline), Endline (after 6 months of baseline)
  this will be measured by the researcher-developed scale
Qualitative self-evaluation attending the project and being a health champion | Endline (after 6 months of baseline)
  Data will be collected through a open qualitative questionnaire (one/two questions will be asked the participants to share their experience for being a health champion and data will be recorded using a voice recorder).
For community people- Change in health literacy score | Midline (after 3 months of baseline), Endline (after 6 months of baseline)
  This will be measured by the European Health literacy Survey Questionnaire short version (HLS-Q12), Bangla version, which is developed by Finbraten, 2018 in English
For community people- Change in awareness and knowledge score | Midline (after 3 months of baseline), Endline (after 6 months of baseline)
  This will be measured by the researcher-developed scale
For community people- Change in health behavior score | Midline (after 3 months of baseline), Endline (after 6 months of baseline)
  This will be measured by the researcher-developed scale

CONTACTS AND LOCATIONS:
Locations (1):
- Begum Ayesha Pilot Girls' High School And College, Dhaka, Dohar, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Will be shared according to correspondence request.